CLINICAL TRIAL: NCT06616519
Title: Multi-center, Open, Parallel, and Randomly Controlled Comparison Between MSENC1 Soft Hydrophilic Contact Lenses and Oxypure Color Soft Hydrophilic Contact Lenses in Their Safety and Efficacy
Brief Title: A Study to Evaluate the Safety and Efficacy of MSENC1 Soft Hydrophilic Contact Lenses and Oxypure Color Soft Hydrophilic Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BenQ Materials Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSENC1 202101
Record Dates: First submitted 2024-09-19; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BenQ Materials MSENCI lenses (Experimental): BenQ Materials Daily disposable contact lens wears for 1 month
  Interventions: Device: BenQ Materials MSENCI soft hydrophilic contact lenses
- Visco Oxypure lens (Active Comparator)
  Interventions: Device: Visco Oxypure Color soft hydrophilic contact lenses

INTERVENTIONS:
Device: BenQ Materials MSENCI soft hydrophilic contact lenses — Test lenses were to be worn for approximately 90 days.
  Arms: BenQ Materials MSENCI lenses
Device: Visco Oxypure Color soft hydrophilic contact lenses — Control lenses were to be worn for approximately 90 days
  Arms: Visco Oxypure lens

SUMMARY:
This project is an open, parallel, randomly controlled, and non-inferiority clinical trial of MSENCI soft hydrophilic contact lenses with Oxypure color soft hydrophilic contact lenses used as the control product.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, no gender limitation;
2. Soft hydrophilic contact lenses worn should be from 0.00D to -12.00D;
3. Subjects should have normal binocular conditions without any abnormality or diseases except for ametropia;
4. The optimal binocular CVA with glasses ≥ 1.0;
5. The astigmatism should be ≤1.5D;
6. Binoculus BUT >5s;
7. should accept follow-ups for at least 90 days and wear the contact lens as required in the protocol;
8. should understand the purpose of the trial, volunteer to attend and sign the Informed Consent Form by the subjects themselves or their legal guardians.

   .

Exclusion Criteria:

1. Patients who suffer from systemic diseases that prohibit contact lens use or receive treatment that may affect the vision or contact lens use;
2. Patients who have worn hard contact lenses within 4 weeks or soft contact lenses within 7 days before being included in the trial;
3. Patients who are allergic to contact lenses or suffer from systemic allergy;
4. Patients who have keratoconus or other cornea irregularity;
5. Patients who always stay at places that are dry, dust-heavy, having volatile chemicals or otherwise affect the use of soft hydrophilic contact lenses;
6. People who are pregnant, during their lactation or prepare for the pregnancy while being included;
7. People who have only a single eye qualified for the trial;
8. People who have attended a clinical trial of medicine or medical devices other than contact lens within 3 months before being included in this trial;
9. People who have attended a clinical trial of medicine or medical devices other than contact lens within 3 months before being included in this trial;
10. Other cases where investigators determine the soft contact lens should not be used or the candidate should be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
efficacy evaluation indexes | after wearing lenses for 7 days
  Binocular CVA with lenses after wearing lenses, The percentage of changes in iris color

SECONDARY OUTCOMES:
Time of Break up time (BUT) | on the day of wearing the lens and wearing lenses for 7 days,30 days and 90 days
  Comparison of BUT time results between the experimental group and control group
Distance Uncorrected visual acuity (UCVA) | on the day of wearing the lens and wearing lenses for 7 days,30 days and 90 days
  Comparison of distance uncorrected visual acuity results between the experimental group and control group
Fitness of the contact | on the day of wearing the lens and wearing lenses for 7 days,30 days and 90 days
  the position of lens on the ocular surface, the coverage, tightness and movability of lens

OTHER OUTCOMES:
efficacy evaluation indexes | on the day of wearing the lens and after wearing lenses for 30 days and 90 days
  Instant iris color change after wearing lenses Binocular CVA with lenses ≥ 1.0

CONTACTS AND LOCATIONS:
Locations (1):
- BenQ Materials Corporation, Taoyuan, China

IPD SHARING:
Plan to Share IPD: No